CLINICAL TRIAL: NCT05300633
Title: Adapting Community Reinforcement Approach and Family Training to Target Substance Use in Early Psychosis Intervention: A Pilot Study of Group Therapy
Brief Title: Community Reinforcement Approach and Family Training for Substance Use in Early Psychosis Intervention
Acronym: CRAFT-EPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 127-2021
Record Dates: First submitted 2022-02-10; First posted 2022-03-29 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Psychosis; Schizophrenia and Related Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Substance Use; Substance Use Disorders
Keywords: Group therapy; Community Reinforcement Approach and Family Training
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Single arm pilot study recruiting family member/concerned significant other participants to receive the intervention and complete outcome measures and identified patients to complete outcome measures only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Family member/concerned significant other
  Interventions: Behavioral: Group-Based Community Reinforcement Approach and Family Training-Early Psychosis Intervention (CRAFT-EPI)

INTERVENTIONS:
Behavioral: Group-Based Community Reinforcement Approach and Family Training-Early Psychosis Intervention (CRAFT-EPI) — Behavioral therapy adapted for families of young people experiencing early psychosis delivered via telemedicine to groups following an individual orientation. Group session topics include self-care, communication, functional analysis, positive reinforcement, treatment engagement, natural consequences, and problem solving. A happiness scale will be completed at each session. Will be provided in the context of an early psychosis intervention program that provides coordinated specialty care to 16- to 29-year-olds experiencing any diagnosis that can manifest as early psychosis.

SUMMARY:
The goal of this pilot feasibility and proof of concept study is to evaluate whether Community Reinforcement and Family Training (CRAFT) as adapted for group delivery in an early psychosis intervention (EPI) program has a clinically significant impact on the concerned significant other (CSO) and Identified patient (IP), and whether a larger, definitive trial is feasible. The intervention aims to improve treatment engagement and reduce distress, as reported by the CSO. To assess feasibility of the intervention for a definitive trial of CRAFT-EPI, the investigators will evaluate recruitment, retention, and assessment completion rates.

DETAILED DESCRIPTION:
Substance use has a major impact on the prevalence and course of early psychosis in young people. Substance use disorders occur in over 40% of people with schizophrenia spectrum disorders. There is increasing evidence to support the fact that cannabis can trigger and worsen psychosis. Young people with psychosis who have comorbid substance use disorders are known to experience worse outcomes, with a three-fold risk of psychosis relapse compared to those without substance use disorders. Current Canadian guidelines recommend integration of substance use treatments in early psychosis intervention programs and specifically suggest integrating addiction-based psychosocial interventions, and involving families in care, but there is limited evidence to support any one specific psychosocial intervention in this population. Studies show that around half of young people with psychosis who use substances significantly reduce their use with the general education and advice provided in early psychosis intervention programs, but it is unclear how programs should intervene to support the other half of clients who continue to struggle.

Community Reinforcement Approach and Family Training (CRAFT) grew out of the understanding that individuals with substance use disorders often struggle with treatment-seeking motivation, whereas their family members are typically highly motivated to get help for them. Having a young person in the family with a substance use disorder can be a very distressing experience, leading to marital and family conflict, physical and verbal abuse, financial problems, and mental health problems for their family members. CRAFT helps family members change the family environment in such a way that a non-substance using lifestyle is more rewarding than one focused on the use of substances. CRAFT aims to improve family members' understanding of addiction, learn about their own behaviors that may unintentionally be promoting substance use, and to modify their own behavior to foster a supportive environment. The ultimate goals are to increase the motivation of the person with the substance use disorder to seek help, and to decrease their substance use. CRAFT teaches family members, who often lack support, how to better take care of themselves and their mental health, and increase their happiness independent of whether their loved one enters substance use treatment.

The efficacy of CRAFT has been demonstrated in multiple research trials, with high rates of individuals with substance use disorders entering treatment. Importantly, the treatment engagement outcomes are effective regardless of the age of the family member or their relationship to the identified patient, and the identified patient's substance of choice. While the therapy is typically provided to families one at a time, it has been adapted to be delivered in groups with equivalent efficacy and the added advantage of reaching more families and built-in peer support.

Families who have completed a basic psychoeducation group at the Centre for Addiction and Mental Health (CAMH) Slaight Centre for Early Intervention (SCEI) and are concerned about their identified patient's substance use will be offered participation in a study of group CRAFT. The intervention has been adapted for early psychosis by Dr. Julie McCarthy at McLean Hospital. It will consist of an individual orientation session, 6 weekly group sessions, and a booster session. Families' satisfaction with this model, changes in their level of stress, quality of life, and other outcomes, and the patients' readiness to change, substance use, and engagement in substance use treatment will be evaluated. Families and patients will complete assessments at baseline, post-intervention, and 12-week follow-up. Families will additionally be invited to participate in a focus group that explores their experience of the intervention.

The goal of this pilot feasibility and proof of concept study is to evaluate whether CRAFT as adapted for group delivery in an EPI program has a clinically significant impact on the family and identified patient, and whether a larger, definitive trial is feasible. This intervention has the potential to fill a major gap in early psychosis intervention, improving outcomes for both youth and families.

ELIGIBILITY:
Inclusion Criteria:

Concerned significant other (CSO)

* Adult (at least 18 years) family member of an identified patient (IP) enrolled in SCEI treatment. The IP should be aged 16-29 years with clinician diagnosis of early psychosis (schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I disorder, major depressive disorder with psychotic features, substance-induced psychotic disorder, or unspecified schizophrenia spectrum and other psychotic disorder). The IP does NOT need to be enrolled in the study in order for the CSO to participate. Up to 2 CSOs associated with the same IP may participate.
* Has completed the program's introductory psychoeducation group
* Concerned about substance use in the IP enrolled in the early psychosis intervention program

Identified patient

* Enrolled in the early psychosis intervention program, aged 16-29 years with clinician diagnosis of early psychosis (schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I disorder, major depressive disorder with psychotic features, substance-induced psychotic disorder, or unspecified schizophrenia spectrum and other psychotic disorder)
* Not currently receiving specialized substance use treatment (i.e. by a clinician other than their NAVIGATE clinicians)

Exclusion Criteria:

Concerned significant other

* Inability to provide informed consent
* Inability to communicate in basic oral and written English.
* There are already 2 CSOs associated with a given IP that are participating in the CRAFT-EPI study.
* Lack of a device for videoconferencing and a secure Wi-Fi connection
* Unwilling to turn camera on for weekly group sessions (except in the case of a poor Wi-Fi connection, or other similar circumstances)

Identified patient

* Does not have a CSO that is enrolled in the CRAFT-EPI study
* Inability to provide informed consent
* Inability to communicate in basic oral and written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Rate of treatment entry for substance use | 18 weeks
  Treatment entry for substance use by the identified patient as reported by their family member (concerned significant other)
Rates of recruitment | Baseline
  Number of family member and identified patient participants who consent to participation
Rates of retention | 18 weeks
  Number of family member participants who complete 6 intervention sessions and booster session
Rates of assessment completion | 18 weeks
  Proportion of assessments completed by consented family members and identified patients, averaged over 3 timepoints

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) total score | Baseline, 6 weeks, 18 weeks
  Symptoms of depression
Happiness Scale total score | Baseline, 6 weeks, 18 weeks
  Experience of happiness
Perceived Stress Scale-14 item total score | Baseline, 6 weeks, 18 weeks
  Experience of stress
Ontario Perception of Care Tool-Mental Health and Addictions section scores | 6 weeks, 18 weeks
  Perceptions of care, satisfaction with the model
Contemplation Ladder total score | Baseline, 6 weeks, 18 weeks
  Readiness to change substance use
National Institute on Drug Abuse (NIDA)-Modified Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) V2.0 total score | Baseline, 6 weeks, 18 weeks
  Substance use
Generalized Anxiety Disorder-7 (GAD-7) total score | Baseline, 6 weeks, 18 weeks
  Symptoms of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Kozloff, MD, SM, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meyers RJ, Miller WR, Hill DE, Tonigan JS. Community reinforcement and family training (CRAFT): engaging unmotivated drug users in treatment. J Subst Abuse. 1998;10(3):291-308. doi: 10.1016/s0899-3289(99)00003-6. PMID 10689661